CLINICAL TRIAL: NCT04739748
Title: Prognostic Biomarkers in Predicting Mortality in Respiratory Patients With Ventilator-Associated Pneumonia
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen Aly Mahmoud Abdel Aleem, lecture in Faculty of medicine,Assiut University, Assiut University
Other Study IDs: IRB17300520
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Red cell distribution width; neutrophil-lymphocyte ratio; Intensive care units; Respiratory
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory ICU patient: patient in RICU that developed ventilator-associated pneumonia
  Interventions: Diagnostic Test: complete blood picture

INTERVENTIONS:
Diagnostic Test: complete blood picture — Measure the red blood cell distribution width (RDW), the neutrophil-lymphocyte ratio (NLR).

SUMMARY:
The aim of this study is to evaluate prognostic efficiency RDW and NLR for mortality prediction in respiratory patients with VAP.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is the most common nosocomial infection. VAP continues to be a leading cause of morbidity and mortality in the nosocomial setting. Red cell distribution width (RDW) and neutrophil-lymphocyte ratio (NLR) are prognostic factors to mortality in different diseases.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory failure needs mechanical ventilator support > 48 hrs. VAP was defined as an acute lower respiratory tract infection in mechanically ventilated patient > 48 hrs with a new or progressing infiltrate on chest radiograph and who met at least two of the following clinical criteria: body temperature >38°C or <36°C with no other recognized cause, white blood cell count >10,000 /mm3 or <5000 /mm3, or a macroscopically purulent tracheal aspirate
* Only the first VAP episode was included

Exclusion Criteria:

* Neutropenia (< 500 cells/ml) before the development of VAP.
* Conditions are known to influence total and differential WBC counts such as chronic inflammatory conditions, hematologic disorders, history of chemotherapy, or radiotherapy within 4 weeks before enrollment.
* Conditions are known to affect RDW as anemia due to nutritional deficiency (ie, iron, vitamin B12, and folic acid).
* Patients with HIV/AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with the clinical suspicion of VAP in the Respiratory ICU were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | 45 days
  The number of patients who not Survive after developing ventilator-associated pneumonia in their stay in the Respiratory Intensive Care Unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Department-faculty of medicine-Assuit university, Asyut, Egypt

REFERENCES:
- [Result] Huang KT, Tseng CC, Fang WF, Lin MC. An early predictor of the outcome of patients with ventilator-associated pneumonia. Chang Gung Med J. 2010 May-Jun;33(3):274-82. PMID 20584505
- [Result] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Result] Bello S, Fandos S, Lasierra AB, Minchole E, Panadero C, Simon AL, Gavin O, De Pablo F, Menendez R, Torres A. Red blood cell distribution width [RDW] and long-term mortality after community-acquired pneumonia. A comparison with proadrenomedullin. Respir Med. 2015 Sep;109(9):1193-206. doi: 10.1016/j.rmed.2015.07.003. Epub 2015 Jul 14. PMID 26205553